CLINICAL TRIAL: NCT06827821
Title: Preliminary Evaluation of the Safety, Pharmacokinetics, and Clinical Application of 18F-CP6A PET Imaging in Synucleinopathies
Brief Title: Application of 18F-CP6A PET Imaging in Synucleinopathies
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Shenzhen Braegen Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-1220
Record Dates: First submitted 2024-12-20; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Synucleinopathies
MeSH Terms: conditions — Synucleinopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET imaging targeting α-synuclein in synucleinopathies (Experimental): Determine if targeting α-synuclein PET is safe and effective method for imaging of synucleinopathies
  Interventions: Drug: 18F-CP6A

INTERVENTIONS:
Drug: 18F-CP6A — For pharmacokinetics, healthy volunteers underwent PET imaging targeting α-synuclein. Blood samples were collected at before and 2 ± 1, 5 ± 2, 10 ± 2, 30 ± 5, 60 ± 5, 90 ± 5, and 120 ± 10 min after imaging agent injection, and urine specimens were collected at before and 0-1.5, and 1.5-3 h after injection to measure radioactivity in blood and urine. PET/MR and PET/CT scans were performed at 0 ± 10, 30 ± 10, 60 ± 10, and 100 ± 10 min after injection to understand distribution for healthy volunteers and synucleinopathy patients. A separate 10-minute PET scan of the brain is required of each acquisition. Blood tests, liver and kidney function, and other biochemical markers must be performed one week prior to and after imaging.

SUMMARY:
Synucleinopathies are a group of severe neurodegenerative diseases, including Parkinson's Disease (PD), Dementia with Lewy Bodies (DLB), and Multiple System Atrophy (MSA). A common feature of these diseases is the pathological aggregation of α-synuclein (α-Syn), which forms Lewy Bodies (LBs), directly causing neuronal damage and death. Clinically, these diseases can present similar parkinsonian syndromes, making differential diagnosis more challenging. However, they may exhibit significant differences in the distribution and morphology of α-Syn pathology. For example, in MSA, the pathological α-Syn primarily accumulates in oligodendrocytes, particularly in the brainstem and cerebellar white matter, which differs significantly from the neuronal Lewy Body formation seen in PD and DLB.

Currently, imaging biomarkers related to β-amyloid (Aβ) and tau proteins have been widely used in clinical diagnosis and research. However, imaging biomarkers targeting α-Syn are still relatively lacking, which limits the early diagnosis and accurate subtyping of these diseases.

In recent years, some PET imaging agents targeting α-Syn have demonstrated good affinity in vitro and in animal experiments, significantly outperforming other common neurodegenerative biomarkers, including Aβ and tau proteins. These agents show promising potential in aiding the diagnosis of synucleinopathies. Professor Ye Keqiang's team at Shenzhen University of Technology has previously developed a small molecule compound (F0502B) with high affinity and selectivity for α-Syn aggregates. Early in vivo and in vitro experiments showed that it could specifically bind to LBs and quantify the amount of LBs in the brain, aiding the early detection of preclinical PD patients and dynamic monitoring of disease progression. Further optimization of the F0502B compound led to the development of its derivative, CP6A. The 18F-labeled probe of CP6A preferentially highlights α-Syn deposition in the brains of animal models and has demonstrated good safety in both mice and monkeys.

Based on the above, this project intends to include clinically diagnosed or highly probable synucleinopathy patients and healthy volunteers, using the 18F-labeled derivative of the α-synuclein-specific imaging agent, 18F-CP6A, to perform integrated PET imaging. The goal is to explore the in vivo safety, pharmacokinetics, and clinical application value of 18F-CP6A in synucleinopathies.

DETAILED DESCRIPTION:
Neurodegenerative diseases represent a significant global health challenge. With the increasing life expectancy, it is estimated that by 2050, the number of individuals suffering from dementia will reach 50 million. Among these diseases, Parkinson's disease (PD) is the second most common neurodegenerative disease, following Alzheimer's disease (AD). The typical pathological features of PD include the loss of dopaminergic neurons and the accumulation of α-synuclein (α-Syn), leading to the formation of Lewy bodies. Other diseases with similar pathological features of α-Syn accumulation include Dementia with Lewy Bodies (DLB) and Multiple System Atrophy (MSA). However, many neurodegenerative diseases, including those related to synucleinopathies, can present with similar parkinsonian syndromes, making differential diagnosis challenging.

α-Synuclein has emerged as a potential diagnostic and differential diagnostic biomarker for synucleinopathies. The deposition of α-Syn is a common characteristic of these diseases, and pathological examinations have shown significant heterogeneity in the deposition patterns across different synucleinopathies. In PD, α-Syn typically appears as intracellular inclusions within neurons, first appearing in the brainstem, then spreading to the midbrain/substantia nigra, and eventually to the medial temporal cortex and neocortex. In DLB, α-Syn distribution is more widespread in cortical regions compared to PD, while in MSA, α-Syn deposits are primarily found in oligodendrocytes, particularly in the white matter of the brainstem and cerebellum. Therefore, in vivo imaging of α-Syn could be an important tool for diagnosing and differentiating synucleinopathies.

Positron emission tomography (PET) has been widely used for diagnosing neurodegenerative diseases, using probes targeting amyloid β (Aβ) and tau proteins for AD. However, the deposition of α-Syn is usually less prominent than that of Aβ and tau. Additionally, dopamine transporter (DAT) and vesicular monoamine transporter type 2 (VMAT2) imaging are also used for diagnosing PD but are less effective for distinguishing atypical Parkinsonism or other conditions affecting the nigrostriatal pathway. These imaging techniques are also highly sensitive to the effects of dopaminergic medications, which can alter the imaging results. To address these challenges, researchers have developed highly selective α-Syn imaging agents, enabling early diagnosis and monitoring of disease progression in synucleinopathies.

This study aims to evaluate the safety, diagnostic potential, pharmacokinetics, and radiation dose of the α-Syn specific imaging agent, 18F-CP6A, in patients diagnosed with PD, MSA, and DLB, as well as healthy volunteers, using integrated PET/MRI imaging. The specific objectives are:

1. Evaluate the safety of a single intravenous dose of 18F-CP6A in participants.
2. Investigate the potential of 18F-CP6A in aiding the diagnosis of different synucleinopathies.
3. Investigate the pharmacokinetics of 18F-CP6A in healthy volunteers.
4. Investigate the radiation dose to the human body after a single intravenous injection of 18F-CP6A in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

1. Fully understand and voluntarily sign the informed consent form.
2. Aged 18-65 years, any gender.
3. Male weight ≥ 50.0 kg, female weight ≥ 45.0 kg; BMI within 19.0-26.0 kg/m2.
4. Non-synucleinopathy, normal motor function, UPDRS score of 0.
5. No history of other neurological or chronic diseases in the last 3 years.
6. No abnormal vital signs or physical examination findings.
7. No pregnancy or lactation, and willing to use effective contraception during the trial period and for 6 months post-study.
8. No participation in other clinical trials within the past month.
9. Able to communicate effectively with the study team and understand and comply with the study requirements.

Synucleinopathy Patients:

1. Ability to sign the informed consent form or by a legal representative.
2. Aged 50-80 years, any gender.
3. Clinically diagnosed or suspected PD, MSA, or DLB based on diagnostic criteria [including China's Parkinson's Disease Diagnosis (2016), MSA Consensus (2022), and DLB Guidelines (2021)].
4. No other neurological diseases, severe chronic diseases, or malignancies.
5. No family history of neurodegenerative diseases or movement disorders.
6. Female participants of childbearing potential must use contraception throughout the study period.

Exclusion Criteria:

Healthy Volunteers:

1. Any severe or unstable medical condition, acute diseases prior to the study.
2. Pregnant or breastfeeding women.
3. Any surgery within the last 6 months that could affect drug absorption, distribution, metabolism, or excretion.
4. Use of any medication (prescription or over-the-counter) within 2 weeks prior to the study.
5. Inability to undergo PET/MRI or PET/CT imaging (e.g., claustrophobia).
6. Participation in studies involving radioactive substances within the last 12 months.
7. Any other factor that may interfere with study results.

Synucleinopathy Patients:

1. Inability or unwillingness to sign the informed consent form.
2. Pregnant or breastfeeding participants.
3. History of other neurological diseases or severe chronic illnesses.
4. Known allergy to α-Syn imaging agents or synthetic excipients.
5. Inability to complete PET/MR or PET/CT imaging.
6. Researcher assesses poor compliance or other conditions that would render participation unsuitable.
7. Major surgery within the last month.
8. Participation in other clinical trials within the last 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-17 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual and standardized uptake values assessment of biodistribution | From enrollment to the end of imaging at 4 weeks
  At least two experienced nuclear medicine physicians will conduct a visual analysis using consensus reading. The standardized uptake value (SUV) of brain and other organs will be measured after a semiquantitative analysis is conducted for each case. The SUV ranges from 0 to infinity, and a higher score means a higher uptake of targeting α-synuclein probe by the tumor, which implies a greater possibility of synucleinopathies.

SECONDARY OUTCOMES:
Radioactivity in the blood and urine samples | From enrollment to the end of imaging at 4 weeks
  Blood samples will be collected at before injection of 18F-CP6A, and 2 ± 1、5 ± 2、10 ± 2、30 ± 5、60 ± 5、90 ± 5、120 ± 10 minutes after injection. Urine samples were collected at before injection of 18F-CP6A, and 0-1.5 and 1.5-3 hours after injection. Radioactivity in the blood and urine samples will be measured by gamma counters.
Radiation doses in healthy subjects | From enrollment to the end of imaging at 4 weeks
  Calculate the radiation equivalent dose (in mSv/MBq) to each organ tissue in healthy subjects, including: brain, heart, liver, spleen, lungs and kidneys, using OLINDA/EXM software.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China